CLINICAL TRIAL: NCT02171949
Title: Randomized, Open and Controlled Clinical Trial for Evaluation of Treatment With Multiple Infusions of Mononuclear Bone Marrow Cells in Patients With Chronic Liver Diseases
Brief Title: Clinical Trial for Evaluation of Treatment With Multiple Infusions of Mononuclear Bone Marrow Cells in Patients With Chronic Liver Diseases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Rafael (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Ricardo Ribeiro dos Santos, PhD, Hospital Sao Rafael
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCL 03/13
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis; Hepatic Cirrhosis
Keywords: Chronic hepatitis; Hepatic cirrhosis
MeSH Terms: conditions — Hepatitis, Chronic; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention)
- Bone marrow mononuclear cell therapy (Active Comparator)
  Interventions: Biological: Infusion of bone marrow mononuclear cells.

INTERVENTIONS:
Biological: Infusion of bone marrow mononuclear cells. — Patients on this group will receive therapy with mononuclear cells. The cells will be diluted on saline and then injected on the hepatic artery through femoral artery puncture.
  Arms: Bone marrow mononuclear cell therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of multiple infusions of mononuclear bone marrow cells in patients with chronic liver diseases.

DETAILED DESCRIPTION:
This is a safety/efficacy phase II, open, randomized, controlled clinical trial, with two arms. The study population will consist of 30 patients with chronic decompensated liver disease (Child-Pugh B or C). The candidates included in the study will be asked to voluntarily participate and sign the written consent.

The patients will be allocated randomly into 2 groups: in group A, the patients will undergo the intervention; and in group B, the patients will be the controls. Patients of both groups will receive clinical follow-up. They will be maintained on drug therapy commonly used in patients with cirrhosis, which may include: spironolactone, furosemide, lactulose, metronidazole, neomycin, analogs of nucleoside / nucleotide in patients with hepatitis B, and vitamin complexes.

All patients included in Group A will undergo cell therapy according to the technique described as follows: on day 1 (D-1), patients will be hospitalized to undergo the bone marrow puncture through the iliac crest. 150 to 200 ml of bone marrow aspirate will be collected. The procedure will be done under local anesthesia and sedation. The fraction of mononuclear cells will be isolated from the aspirated marrow by the SEPAX (System of cell processing) - Biosafe, Switzerland.

The enriched fraction of collected mononuclear cells will be resuspended in saline. The obtained cell populations will be analyzed by flow cytometry for its characterization, and then diluted in 20 ml saline. The cells will be injected 3 times throughout the study, on days 1 (D-1), 30 (D-30) and 60 (D-60).

Patients will undergo a series of clinical and laboratory evaluations and will also be submitted to the following procedures:

* Cell blood count
* Biochemical analysis (measurement of electrolytes - sodium and potassium)
* Renal function tests (urea and creatinine)
* Liver profile tests (total proteins and fractions, bilirubin, prothrombin time, transaminases, alkaline phosphatase, gamma-GT)
* Metabolic profile (glucose, total cholesterol and fractions, triglycerides)
* Thyroid profile tests
* Serology required for blood transfusion and bone marrow transplant in Brazil
* Alpha-fetoprotein
* Beta-HCG (human chorionic gonadotropin), for women
* Handgrip dynamometer
* Treadmill test
* Six-minute walk test
* Abdomen doppler ultrasound
* Magnetic resonance imaging of the upper abdomen with elastography
* Measurement of serum factors
* Shear wave elastography

Also, the patients will respond to questions from the SF (Short Form) -36 questionnaire (for assessment of quality of life).

Clinical follow-up will be kept for patients who suspend their participation in the study for any adverse event and / or laboratory abnormality, or for the patient's own desire, following insurance protocols. In addition to the clinical and surgical follow-up, specific medical care will be offered to patients who experience adverse events, until stabilization of the patient, even if the target date for completion of the study has been exceeded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis of different etiologies, confirmed by clinical examination, laboratory tests, imaging studies and / or biopsy that shows process of evolution to cirrhosis or established cirrhosis (equivalent to Metavir score F3/F4);
* Non-participation on the waiting list for liver transplantation or, in case of participation, allocation after the fifth position in the list, for subjects with blood group A or O, and after the third position for subjects with other blood groups;
* Absence of clinical, laboratory and radiological evidence of hepatocellular carcinoma;
* Absence of pregnancy potential or negative pregnancy test for female patients, or impossibility to use a contraception method during the study;
* Permission for doing the puncture of iliac crest after evaluation of pre-anesthetic visit.

Exclusion Criteria:

* Impossibility to obtain vascular access for percutaneous procedure;
* Sepsis;
* Hepatic encephalopathy detected at the screening tests;
* Budd-Chiari syndrome;
* Severe coagulopathy with INR > 2,4 or platelet count < 30.000;
* Presence of malignancies (excluding non-melanoma skin cancer);
* Decompensated heart failure;
* Primary hematologic diseases;
* Renal failure with creatinin > 2,5mg/dl;
* Coinfection with HIV;
* Pregnancy;
* Dependence of organic medium such as circulatory or ventilatory;
* Any other comorbidity with an impact on the survival in 2 years;
* Participation in other clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Child-Pugh score | 12 months
  Functional class improvement of 2 points on Child-Pugh score.
Evaluation of MELD score | 12 months
  Functional class improvement of 2 points on MELD score.

SECONDARY OUTCOMES:
Degree of muscle strength | 12 months
  Improvement in the degree of muscle strength assessed using handgrip dynamometer.
Hepatic fibrosis | 12 months
  Decrease of hepatic fibrosis detected by elastography shear waves.
Quality of life | 12 months
  Improvement on the SF-36 questionnaire score, which evaluates quality of life.
Evaluation of functional capacity | 12 months
  Improvement in the functional capacity, assessed by six-minute walk test.
Evaluation of serum bilirubin levels | 12 months
  Improvement in the serum bilirubin levels.
Evaluation of serum albumin levels | 12 months
  Improvement in the serum albumin levels.
Evaluation of prothrombin time | 12 months
  Improvement in prothrombin time.
Evaluation of serum levels of cytokines | 12 months
  Decrease in the serum levels of cytokines.
Evaluation of fibrosis markers levels | 12 months
  Decrease in the serum levels of fibrosis markers.

CONTACTS AND LOCATIONS:
Overall Officials: André C Lyra, PhD, Principal Investigator — Hospital São Rafael; Bruno SF Souza, MD, Msc, Study Chair — Hospital São Rafael; Eduardo L Braga, PhD, Study Chair — Hospital São Rafael; Lourianne N Cavalcante, PhD, Study Chair — Hospital São Rafael; Milena BP Soares, PhD, Study Chair — Hospital São Rafael; Ricardo R dos Santos, PhD, Principal Investigator — Hospital São Rafael; Ticiana F Larocca, MD, Msc, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil